CLINICAL TRIAL: NCT06797245
Title: The APPROVE Trial: A Randomized Controlled Trial Evaluating the Efficacy and Safety of a Prescription Digital Therapeutic for Treatment of Overactive Bladder in Women
Brief Title: APPROVE Trial: Evaluating a Prescription Digital Therapeutic for Treatment of OAB in Women
Acronym: APPROVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Foundation for Female Health Awareness (FFHA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APPROVE
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-06

CONDITIONS: Overactive Bladder (OAB); Urinary Urgency; Urinary Urge Incontinence (UUI); Nocturia; Urinary Frequency
Keywords: Overactive Bladder (OAB)
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Nocturia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - RiSolve PDTx App (Experimental): Participants randomized to intervention will be given access to the RiSolve PDTx app for 10 weeks after initial activation.
  Interventions: Device: RiSolve App
- Control - Standard Therapy (Active Comparator): Participants randomized to the control will receive a brief explanation of behavioral therapy with details provided in the form educational handouts including the American Urogynecologic Society (AUGS) "Overactive Bladder" and "Pelvic Floor Muscles and Bladder Training" Patient Fact Sheets.
  Interventions: Behavioral: AUGS Patient Handouts

INTERVENTIONS:
Device: RiSolve App — Participants randomized to intervention will be given access to the RiSolve PDTx app for 10 weeks after initial activation.
  Arms: Intervention - RiSolve PDTx App
Behavioral: AUGS Patient Handouts — AUGS "Overactive Bladder" and "Pelvic Floor Muscles and Bladder Training" Patient Fact Sheets will be provided and reviewed.
  Arms: Control - Standard Therapy

SUMMARY:
The APPROVE trial is a multi-centered, randomized controlled trial designed to assess differences in symptom improvement, quality of life, bladder symptoms, satisfaction with treatment and continued treatment efficacy in women with overactive bladder (OAB) randomized to a prescription digital therapeutic (PDTx) app called RiSolve compared to standard behavioral education (handouts).

DETAILED DESCRIPTION:
In this trial, we will employ a randomized controlled trial design to determine if women with overactive bladder (OAB) treated with the RiSolve prescription digital therapeutic (PDTx) demonstrate greater improvement in OAB-related health as compared to standard behavioral education with informational handouts. RiSolve is a digital therapeutic device intended to provide behavioral therapy and cognitive behavioral therapy (CBT) for adult women who have been diagnosed with OAB, which includes urinary urgency with or without urge urinary incontinence (UUI), urinary frequency, nocturia, and mixed incontinence with predominant OAB symptoms. RiSolve is indicated as an 8-week treatment to reduce the symptoms of OAB.

For the purposes of this trial, the primary outcome to determine improvement in OAB-related health will be defined as achieving the MID (defined as an improvement of 10 points or more) on the OAB-q SF Symptom Severity subscale after 8 weeks of treatment. Secondary outcomes will include achieving the MID on the OAB-q SF Health-Related Quality of Life subscale, meeting the patient's acceptable symptoms state (PASS) on the Patient Global Impression of Severity (PGI-S) and Patient Global Impression of Improvement (PGI-I), and improvements in frequency, nocturia and urge urinary incontinence (UUI) on a 3-day bladder diary and on the ICIQ-FLUTS. Participants will be randomized to either PDTx therapy (active) or standard treatment of behavioral education (control). Participants randomized to control will have the option to crossover to PDTx after the initial 8 weeks of the trial if desired. Participants will continue to be followed and asked about their symptoms at 6 and 12 months.

The impact of this trial has enormous potential to improve treatment of OAB. The ability to offer behavioral therapy via PDTx will reduce patient burden while simultaneously increasing quality of life for women suffering from OAB and decreasing provider burden. The high-quality data from this study will be used to support a marketing application with the FDA through the De Novo pathway for an accessible, low-burden, efficient intervention to help millions of women currently suffering from this burdensome condition.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 22 years old
* Bothersome OAB symptoms (defined as bother rating ≥ 5 on ICIQ-FLUTS question #3b or #9b)
* English-speaking
* Willing to forego other treatment outside of medications for the 8-week trial period
* Use of at least one mobile App

Exclusion Criteria:

* Stress-predominant mixed urinary incontinence (defined as QUID stress score > QUID urge score)
* Voiding dysfunction defined as response ≥ 2 on ICIQ-FLUTS question #7a
* Bladder pain defined as response ≥ 2 on ICIQ-FLUTS question #4a
* Use of an OAB medication (anticholinergic or beta-agonist) within the past two weeks
* Currently using intermittent or indwelling catheter
* History of bladder/urethral, colon/anal, or cervical cancer
* Current or prior use of sacral neuromodulation, tibial stimulation or onabotulinum toxin type A intradetrusor injection
* Currently taking antibiotics/drugs for urinary tract infection^
* Currently undergoing or unwilling to forego pelvic floor physical therapy with a physical therapist or prescription device for the 8-week intervention period
* Planning surgery for pelvic organ prolapse within 12 months of randomization
* Pelvic surgery within the past 6 months
* Planning to undergo pessary fitting °

  * Those on antibiotics for urinary tract infection will be eligible for enrollment 2 weeks after completing antibiotic therapy with subjective resolution of UTI symptoms °Will be eligible after completing pessary fitting

https://researchdata.medstar.net/redcap/surveys/?s=MM7WN7EXACX4PNXJ

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Overactive Bladder Questionnaire short-form (OAB-q SF) | 8 Weeks
  The OAB-q SF is utilized to assess the impact of OAB symptoms on the patient's life,35 and has been shown to be responsive to reductions in urinary urgency, frequency and incontinence during anticholinergic therapy.3 The scale ranges from 0 to 100 with a higher score indicating worse symptom severity. The MID is defined as a change of 10 points

SECONDARY OUTCOMES:
OAB-q SF Health-Related Quality of Life (HRQL) | 8 Weeks
  The OAB-q SF Health-Related Quality of Life (HRQL) subscale is a13-item health-related quality of life subscale of the OAB-q SF. The scale ranges from 0 to 100 with a higher score indicating better quality of life. The MID is defined as a change of 10 points.
Patient Global Impression of Severity (PGI-S) | 8 Weeks
  Patient Global Impression of Severity (PGI-S) is a single item questionnaire to assess a person's impression of disease severity. For purposes of this trial, it will ask participants to "Check the one number that best describes how your urinary tract condition is now" on a 4-point Likert scale ranging from (1) "normal" to (4) "severe". The PASS threshold PGI-S score is < 3.
Patient Global Impression of Improvement (PGI-I) | 8 Weeks
  The Patient Global Impression of Improvement (PGI-I) is a single item questionnaire to assess an individual's impression of change in urinary symptoms. For purposes of this trial the PGI-S has been adapted by removing "taking medication" and it will ask participants to "Check the one number that best describes how your urinary tract condition is now, compared with how it was before you began this study" on a 7-point Likert scale ranging from (1) "very much better" to (7) "very much worse". The PASS threshold PGI-I score is < 3.
3-Day Bladder Diary | 8 Weeks
  A 3-day Bladder Diary will be an electronic bladder diary collected over a 3-day (72 hour) period focusing specifically on number of voids per day, number of voids per night, and number of urinary incontinence (UI) episodes and whether these events are associated with urgency.
Questionnaire for Urinary Incontinence Diagnosis (QUID) | 8 Weeks
  The Questionnaire for Urinary Incontinence Diagnosis (QUID) is a 6-item UI symptom questionnaire to distinguish stress and urgency UI. The QUID serves both as a diagnostic tool to assess UI type and as a measure of SUI and UUI frequency before and after treatment. Prior research has shown that a cut off QUID stress score ≥ 4 and QUID urge score ≥ 6 identify UI type (SUI, UUI or mixed) accurately in 80% of patients as compared to provider diagnosis.
International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) | 8 Weeks
  The International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) is a 12-item questionnaire to evaluate female lower urinary tract symptoms and impact on quality of life derived from the BFLUTS-SF questionnaire. The ICIQ-FLUTS asks each person to rate the frequency of a specific lower urinary tract symptom (such as urgency, frequency, nocturia, nocturnal enuresis, stress incontinence, pain, etc.) on various 5 point scales and then asks the participant to rate the level of bother from that specific symptom on a Likert scale from (0) "not at all" to (10) "a great deal".
Short Personal Experience Questionnaire (SPEQ) | 8 Weeks
  The Short Personal Experience Questionnaire (SPEQ) is a 13-item questionnaire that assesses sexual enjoyment, desire, arousal, orgasm, dyspareunia, sexual activity, sexual partner, and partner limitations. To limit participant burden, the SPEQ has been modified to a shorter 8-item version to include fewer items on partner limitations.
Mobile Application Rating Scale: user version (uMARS) | 8 Weeks
  The Mobile Application Rating Scale: user version (uMARS) is comprised of a 20-item objective quality rating with 4 subscales (engagement, functionality, aesthetics, and information quality), and 6-item subjective quality rating. Higher scores are more desirable. Participants randomized to or who crossover to PDTx treatment will be asked to complete the uMARS questionnaire 8 weeks after starting PDTx treatment. A uMARS score of ≥ 3 is considered acceptable.
Treatment Satisfaction | 8 Weeks
  Treatment satisfaction will be assessed by asking participants to "Rate your level of satisfaction with the study treatment" they received on a 5-point Likert scale ranging from (1) "very satisfied" to (5) "very dissatisfied".
Treatment accessibility | 8 Weeks
  Treatment accessibility will be assessed by recording the number of participants who are unable to or have difficulty accessing the App and any phone calls/tech support requests.
Treatment adherence | 8 Weeks
  Treatment adherence for participants receiving PDTx treatment will be assessed via App usage data. For the control group direct questioning will be used to assess treatment adherence (Did you read the leaflet? Answer choices: Yes / No. If yes, how much of it did you read? With answer choices in % categories; If yes, did you return to the leaflet during the 8 weeks to refresh your memory? Answer choices: Yes / No). For those prescribed an anticholinergic or beta-agonist medication we will assess medication compliance through direct patient questioning to assess if the medication was obtained from the pharmacy, how long the medication was taken, any side effects, and, if applicable, the reason for stopping the medication.
Other Treatments | 12 Months
  Other treatments will be assessed following the initial 8-week intervention period by querying participants as to whether they have any new conditions or are using or have tried using additional treatments that could affect OAB symptoms. These will include assessing for diagnosis of and treatment for stress urinary incontinence, urinary retention, pelvic organ prolapse, genitourinary syndrome of menopause, vaginal atrophy, pregnancy, sleep apnea, heart failure, and diabetes.
Adverse Events | 12 Months
  Adverse events will be assessed by querying participants regarding any adverse events that may occur throughout the trial

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - MedStar Health, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Curavit, Boston, Massachusetts
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Allegheny Health, Pittsburgh, Pennsylvania
  - Medical University of South Carolina Health, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Participant data will be collected and analyzed as an aggregate for any results.

REFERENCES:
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Obstet Gynecol. 2010 May;115(5):1063-1070. doi: 10.1097/AOG.0b013e3181d9d421. No abstract available. PMID 20410783
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Rubin D. Multiple Imputation for Nonresponse in Surveys. New York: John Wiley & Sons, Inc.; 1987.
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Coyne KS, Thompson CL, Lai JS, Sexton CC. An overactive bladder symptom and health-related quality of life short-form: validation of the OAB-q SF. Neurourol Urodyn. 2015 Mar;34(3):255-63. doi: 10.1002/nau.22559. Epub 2014 Jan 13. PMID 25783168
- [Background] Burkett LS, Siddique M, Zeymo A, Brunn EA, Gutman RE, Park AJ, Iglesia CB. Clobetasol Compared With Fractionated Carbon Dioxide Laser for Lichen Sclerosus: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jun 1;137(6):968-978. doi: 10.1097/AOG.0000000000004332. PMID 33957642
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Wilson H. Development and Validation of the User Version of the Mobile Application Rating Scale (uMARS). JMIR Mhealth Uhealth. 2016 Jun 10;4(2):e72. doi: 10.2196/mhealth.5849. PMID 27287964
- [Background] Dennerstein L, Lehert P, Dudley E. Short scale to measure female sexuality: adapted from McCoy Female Sexuality Questionnaire. J Sex Marital Ther. 2001 Jul-Sep;27(4):339-51. doi: 10.1080/009262301317081098. PMID 11441518
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Brookes ST, Donovan JL, Wright M, Jackson S, Abrams P. A scored form of the Bristol Female Lower Urinary Tract Symptoms questionnaire: data from a randomized controlled trial of surgery for women with stress incontinence. Am J Obstet Gynecol. 2004 Jul;191(1):73-82. doi: 10.1016/j.ajog.2003.12.027. PMID 15295345
- [Background] Bradley CS, Rovner ES, Morgan MA, Berlin M, Novi JM, Shea JA, Arya LA. A new questionnaire for urinary incontinence diagnosis in women: development and testing. Am J Obstet Gynecol. 2005 Jan;192(1):66-73. doi: 10.1016/j.ajog.2004.07.037. PMID 15672005
- [Background] Bradley CS, Rahn DD, Nygaard IE, Barber MD, Nager CW, Kenton KS, Siddiqui NY, Abel RB, Spino C, Richter HE. The questionnaire for urinary incontinence diagnosis (QUID): validity and responsiveness to change in women undergoing non-surgical therapies for treatment of stress predominant urinary incontinence. Neurourol Urodyn. 2010 Jun;29(5):727-34. doi: 10.1002/nau.20818. PMID 19787711
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Background] Coyne K, Revicki D, Hunt T, Corey R, Stewart W, Bentkover J, Kurth H, Abrams P. Psychometric validation of an overactive bladder symptom and health-related quality of life questionnaire: the OAB-q. Qual Life Res. 2002 Sep;11(6):563-74. doi: 10.1023/a:1016370925601. PMID 12206577
- [Background] Sanderson DJ, Zavez A, Meekins AR, Eddib A, Lee TG, Barber MD, Duecy E. The Patient Acceptable Symptom State in Female Urinary Incontinence. Female Pelvic Med Reconstr Surg. 2022 Jan 1;28(1):33-39. doi: 10.1097/SPV.0000000000001055. PMID 34009829
- [Background] Funada S, Watanabe N, Goto T, Negoro H, Akamatsu S, Uozumi R, Kishimoto S, Ichioka K, Segawa T, Furukawa TA, Ogawa O. Clinical feasibility and acceptability of adding cognitive behavioral therapy to pharmacotherapy for drug-resistant overactive bladder in women: A single-arm pilot study. Low Urin Tract Symptoms. 2021 Jan;13(1):69-78. doi: 10.1111/luts.12333. Epub 2020 Jul 3. PMID 32618414
- [Background] Price JR, Mitchell E, Tidy E, Hunot V. Cognitive behaviour therapy for chronic fatigue syndrome in adults. Cochrane Database Syst Rev. 2008 Jul 16;2008(3):CD001027. doi: 10.1002/14651858.CD001027.pub2. PMID 18646067
- [Background] Laird KT, Tanner-Smith EE, Russell AC, Hollon SD, Walker LS. Short-term and Long-term Efficacy of Psychological Therapies for Irritable Bowel Syndrome: A Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2016 Jul;14(7):937-947.e4. doi: 10.1016/j.cgh.2015.11.020. Epub 2015 Dec 22. PMID 26721342
- [Background] Glombiewski JA, Sawyer AT, Gutermann J, Koenig K, Rief W, Hofmann SG. Psychological treatments for fibromyalgia: a meta-analysis. Pain. 2010 Nov;151(2):280-295. doi: 10.1016/j.pain.2010.06.011. Epub 2010 Aug 19. PMID 20727679
- [Background] Luo C, Sanger N, Singhal N, Pattrick K, Shams I, Shahid H, Hoang P, Schmidt J, Lee J, Haber S, Puckering M, Buchanan N, Lee P, Ng K, Sun S, Kheyson S, Chung DC, Sanger S, Thabane L, Samaan Z. A comparison of electronically-delivered and face to face cognitive behavioural therapies in depressive disorders: A systematic review and meta-analysis. EClinicalMedicine. 2020 Jun 27;24:100442. doi: 10.1016/j.eclinm.2020.100442. eCollection 2020 Jul. PMID 32775969
- [Background] Hanlon I, Hewitt C, Bell K, Phillips A, Mikocka-Walus A. Systematic review with meta-analysis: online psychological interventions for mental and physical health outcomes in gastrointestinal disorders including irritable bowel syndrome and inflammatory bowel disease. Aliment Pharmacol Ther. 2018 Aug;48(3):244-259. doi: 10.1111/apt.14840. Epub 2018 Jun 14. PMID 29901820
- [Background] Etzelmueller A, Vis C, Karyotaki E, Baumeister H, Titov N, Berking M, Cuijpers P, Riper H, Ebert DD. Effects of Internet-Based Cognitive Behavioral Therapy in Routine Care for Adults in Treatment for Depression and Anxiety: Systematic Review and Meta-Analysis. J Med Internet Res. 2020 Aug 31;22(8):e18100. doi: 10.2196/18100. PMID 32865497
- [Background] Melotti IGR, Juliato CRT, Tanaka M, Riccetto CLZ. Severe depression and anxiety in women with overactive bladder. Neurourol Urodyn. 2018 Jan;37(1):223-228. doi: 10.1002/nau.23277. Epub 2017 Apr 13. PMID 28407347
- [Background] Melotti IGR, Juliato CRT, Coelho SCA, Lima M, Riccetto CLZ. Is There Any Difference Between Depression and Anxiety in Overactive Bladder According to Sex? A Systematic Review and Meta-Analysis. Int Neurourol J. 2017 Sep;21(3):204-211. doi: 10.5213/inj.1734890.445. Epub 2017 Sep 12. PMID 28954462
- [Background] Lai HH, Shen B, Rawal A, Vetter J. The relationship between depression and overactive bladder/urinary incontinence symptoms in the clinical OAB population. BMC Urol. 2016 Oct 6;16(1):60. doi: 10.1186/s12894-016-0179-x. PMID 27716241
- [Background] Harvey J, Finney S, Stewart L, Gillespie J. The relationship between cognition and sensation in determining when and where to void: the concept of cognitive voiding. BJU Int. 2012 Dec;110(11):1756-61. doi: 10.1111/j.1464-410X.2012.11078.x. Epub 2012 May 29. PMID 22642959
- [Background] Sooknarine C, Farrell S, Sarma S, Salameh F, Burke N, Staunton B, Carr E, Sexton K, Agnew G, Downey A, D'Arcy F, Cundiff GW. Pilot Study of a Digital Behavioral Therapy for Overactive Bladder in Women. Urogynecology (Phila). 2024 Dec 1;30(12):956-961. doi: 10.1097/SPV.0000000000001499. Epub 2024 May 7. PMID 38465995
- [Background] Lightner DJ, Gomelsky A, Souter L, Vasavada SP. Diagnosis and Treatment of Overactive Bladder (Non-Neurogenic) in Adults: AUA/SUFU Guideline Amendment 2019. J Urol. 2019 Sep;202(3):558-563. doi: 10.1097/JU.0000000000000309. Epub 2019 Aug 8. PMID 31039103
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Gormley EA, Lightner DJ, Faraday M, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline amendment. J Urol. 2015 May;193(5):1572-80. doi: 10.1016/j.juro.2015.01.087. Epub 2015 Jan 23. PMID 25623739
- [Background] Olivera CK, Meriwether K, El-Nashar S, Grimes CL, Chen CC, Orejuela F, Antosh D, Gleason J, Kim-Fine S, Wheeler T, McFadden B, Balk EM, Murphy M; Systematic Review Group for the Society of Gynecological Surgeons. Nonantimuscarinic treatment for overactive bladder: a systematic review. Am J Obstet Gynecol. 2016 Jul;215(1):34-57. doi: 10.1016/j.ajog.2016.01.156. Epub 2016 Feb 4. PMID 26851599
- [Background] Hu TW, Wagner TH, Bentkover JD, Leblanc K, Zhou SZ, Hunt T. Costs of urinary incontinence and overactive bladder in the United States: a comparative study. Urology. 2004 Mar;63(3):461-5. doi: 10.1016/j.urology.2003.10.037. PMID 15028438
- [Background] Chermansky CJ, Chancellor MB. Increasing awareness and improving the care of urinary incontinence: highlights from the world health organization 2nd international consultation on incontinence july 1-4, 2001, paris, france. Rev Urol. 2003 Winter;5(1):22-5. No abstract available. PMID 16985613
- [Background] Wadensten T, Nystrom E, Nord A, Lindam A, Sjostrom M, Samuelsson E. App-based self-management of urgency and mixed urinary incontinence in women: One-year follow-up. Neurourol Urodyn. 2022 Apr;41(4):945-954. doi: 10.1002/nau.24898. Epub 2022 Mar 9. PMID 35266189
- [Background] Liberman JN, Hunt TL, Stewart WF, Wein A, Zhou Z, Herzog AR, Lipton RB, Diokno AC. Health-related quality of life among adults with symptoms of overactive bladder: results from a U.S. community-based survey. Urology. 2001 Jun;57(6):1044-50. doi: 10.1016/s0090-4295(01)00986-4. PMID 11377301
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Shamliyan T, Wyman J, Bliss DZ, Kane RL, Wilt TJ. Prevention of urinary and fecal incontinence in adults. Evid Rep Technol Assess (Full Rep). 2007 Dec;(161):1-379. PMID 18457475
- [Background] Hagglund D, Walker-Engstrom ML, Larsson G, Leppert J. Quality of life and seeking help in women with urinary incontinence. Acta Obstet Gynecol Scand. 2001 Nov;80(11):1051-5. PMID 11703207
- [Background] Coyne KS, Zhou Z, Thompson C, Versi E. The impact on health-related quality of life of stress, urge and mixed urinary incontinence. BJU Int. 2003 Nov;92(7):731-5. doi: 10.1046/j.1464-410x.2003.04463.x. PMID 14616456
- [Background] Coyne KS, Sexton CC, Irwin DE, Kopp ZS, Kelleher CJ, Milsom I. The impact of overactive bladder, incontinence and other lower urinary tract symptoms on quality of life, work productivity, sexuality and emotional well-being in men and women: results from the EPIC study. BJU Int. 2008 Jun;101(11):1388-95. doi: 10.1111/j.1464-410X.2008.07601.x. PMID 18454794
- [Background] Chiaffarino F, Parazzini F, Lavezzari M, Giambanco V; Gruppo Interdisciplinare di Studio Incontinenza Urinaria (GISIU). Impact of urinary incontinence and overactive bladder on quality of life. Eur Urol. 2003 May;43(5):535-8. doi: 10.1016/s0302-2838(03)00097-6. PMID 12705999
- [Background] Abrams P, Kelleher CJ, Kerr LA, Rogers RG. Overactive bladder significantly affects quality of life. Am J Manag Care. 2000 Jul;6(11 Suppl):S580-90. PMID 11183901
- [Background] Coyne KS, Matza LS, Thompson CL, Kopp ZS, Khullar V. Determining the importance of change in the overactive bladder questionnaire. J Urol. 2006 Aug;176(2):627-32; discussion 632. doi: 10.1016/j.juro.2006.03.088. PMID 16813906
- [Background] Matza LS, Thompson CL, Krasnow J, Brewster-Jordan J, Zyczynski T, Coyne KS. Test-retest reliability of four questionnaires for patients with overactive bladder: the overactive bladder questionnaire (OAB-q), patient perception of bladder condition (PPBC), urgency questionnaire (UQ), and the primary OAB symptom questionnaire (POSQ). Neurourol Urodyn. 2005;24(3):215-25. doi: 10.1002/nau.20110. PMID 15747340
- [Background] Coyne KS, Matza LS, Thompson CL. The responsiveness of the Overactive Bladder Questionnaire (OAB-q). Qual Life Res. 2005 Apr;14(3):849-55. doi: 10.1007/s11136-004-0706-1. PMID 16022077
- [Background] Wu EQ, Birnbaum H, Marynchenko M, Mareva M, Williamson T, Mallett D. Employees with overactive bladder: work loss burden. J Occup Environ Med. 2005 May;47(5):439-46. doi: 10.1097/01.jom.0000161744.21780.c1. PMID 15891521
- [Background] Dmochowski RR, Newman DK. Impact of overactive bladder on women in the United States: results of a national survey. Curr Med Res Opin. 2007 Jan;23(1):65-76. doi: 10.1185/030079907X159533. PMID 17257467